CLINICAL TRIAL: NCT03314935
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of INCB001158 in Combination With Chemotherapy, in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1/2 Study of INCB001158 in Combination With Chemotherapy in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 01158-203; 2017-002904-29 (EudraCT Number)
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer (BTC); Colorectal Cancer (CRC); Endometrial Cancer; Gastroesophageal Cancer (GC); Ovarian Cancer; Solid Tumors
Keywords: INCB001158; arginase inhibitor; oxaliplatin; leucovorin; 5 fluorouracil; gemcitabine; cisplatin; paclitaxel; solid tumors; colorectal cancer; biliary tract cancer; gastroesophageal cancer; endometrial cancer; ovarian cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Gemcitabine; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Experimental): INCB001158 + FOLFOX
  Interventions: Drug: INCB001158; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- Treatment Group B (Experimental): INCB001158 + gemcitabine/cisplatin
  Interventions: Drug: INCB001158; Drug: Gemcitabine; Drug: Cisplatin
- Treatment Group C (Experimental): INCB001158 + paclitaxel
  Interventions: Drug: INCB001158; Drug: Paclitaxel

INTERVENTIONS:
Drug: INCB001158 — Phase 1: INCB001158 administered orally twice daily at the protocol-defined dose. Phase 2: INCB001158 administered orally twice daily at the recommended dose from Phase 1.
  Other Names: Arginase inhibitor
Drug: Oxaliplatin — Oxaliplatin administered intravenously at the protocol-defined dose and schedule.
  Arms: Treatment Group A
Drug: Leucovorin — Leucovorin at the protocol-defined dose and regimen.
  Arms: Treatment Group A
Drug: 5-Fluorouracil — 5-Fluorouracil at the protocol-defined dose and regimen.
  Arms: Treatment Group A
Drug: Gemcitabine — Gemcitabine at the protocol-defined dose and regimen.
  Arms: Treatment Group B
Drug: Cisplatin — Cisplatin at the protocol-defined dose and regimen.
  Arms: Treatment Group B
Drug: Paclitaxel — Paclitaxel at the protocol-defined dose and regimen.
  Arms: Treatment Group C

SUMMARY:
The purpose of this open-label nonrandomized Phase 1/2 study is to evaluate INCB001158 in combination with chemotherapy in participants with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of selected advanced or metastatic solid tumors.
* Presence of measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Baseline archival tumor specimen available or willingness to undergo a pretreatment tumor biopsy to obtain the specimen.
* Resolution of treatment-related toxicities.
* Adequate hepatic, renal, cardiac, and hematologic function.
* Additional cohort-specific criteria may apply.

Exclusion Criteria:

* Subjects who participated in any other study in which receipt of an investigational study drug or device occurred within 28 days or 5 half-lives (whichever is longer) prior to first dose.
* Has received a prior monoclonal antibody within 4 weeks or 5 half-lives (whichever is shorter) before administration of study drug.
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks before administration of study treatment.
* Has received prior approved radiotherapy within 14 days of study therapy.
* Has had known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has an active infection requiring systemic therapy.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (10):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - USA Mitchell Cancer Center, Mobile, Alabama
  - UC Davis - Comprehensive Cancer Centre, Sacramento, California
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
- Belgium (2):
  - Grand Hopital de Charleroi - Department of Medical Oncology, Brussels
  - Institut Jules Bordet - Clinical Trials Conduct Unit, Brussels
- United Kingdom (2):
  - UCL Cancer Institute, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 11 study centers in the United States, the United Kingdom, and Belgium.
Groups:
- Phase 1: INCB001158 50 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 milligrams (mg) twice daily (BID) starting on Day 1 of each 28-day cycle. Participants also received intravenous modified FOLFOX6 (mFOLFOX6: oxaliplatin 85 mg/meters squared [m^2], leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1: INCB001158 75 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1: INCB001158 100 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle.
- Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle.
- Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle.
- Phase 1: INCB001158 50 mg + Paclitaxel: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 1: INCB001158 75 mg + Paclitaxel: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 1: INCB001158 100 mg + Paclitaxel: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1): In Phase 2, participants with microsatellite-stable-colorectal cancer (MSS-CRC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1): In Phase 2, participants with biliary tract cancer (BTC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 25 mg/m^2 on Day 1 and 8 of each 28-day cycle.
- Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2): In Phase 2, participants with ovarian cancer (OC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 750 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and 8 of each 28-day cycle.
- Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1): In Phase 2, participants with gastroesophageal cancer (GC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2): In Phase 2, participants with endometrial cancer (EC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3): In Phase 2, participants with ovarian cancer (OC) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
Period: Phase 1
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Started | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 2 | 5 | 4 | 3 | 4 | 5 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Captured as "Other" in Database | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 33 | 9 | 11 | 10 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 33 | 9 | 11 | 10 | 24
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 20 | 6 | 7 | 6 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1 | 4 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: INCB001158 100 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cyce after administration of INCB001158.
- Total: Total of all reporting groups
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3) | Total
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7 | 8 | 33 | 9 | 11 | 10 | 24 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.80) | 60.3 (9.93) | 65.2 (7.99) | 54.0 (18.93) | 64.5 (16.82) | 54.0 (15.64) | 62.0 (14.57) | 47.4 (10.29) | 61.4 (6.95) | 62.8 (11.26) | 59.3 (12.74) | 65.3 (8.87) | 58.8 (11.90) | 62.3 (9.29) | 60.6 (9.04) | 59.93 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 3 | 2 | 3 | 5 | 4 | 5 | 3 | 21 | 9 | 4 | 10 | 24 | 103
  Male | 5 | 2 | 3 | 4 | 2 | 1 | 2 | 1 | 2 | 5 | 12 | 0 | 7 | 0 | 0 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 6
  Not Hispanic or Latino | 5 | 5 | 6 | 6 | 4 | 4 | 7 | 5 | 7 | 7 | 29 | 7 | 11 | 10 | 23 | 136
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 6 | 6 | 6 | 3 | 4 | 7 | 5 | 5 | 7 | 31 | 8 | 8 | 8 | 23 | 129
  Black/African-American | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 6
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 7
  American-Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  East Indian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Provided/Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Black/Carribean | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Captured as Hispanic/Latino in Database | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phases 1 and 2: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 1385 days
Population: Full Analysis Set (FAS): all participants enrolled in the study who received at least 1 dose of INCB001158, mFOLFOX6, gemcitabine/cisplatin, or paclitaxel. As pre-defined in the Statistical Analysis Plan, data analysis was conducted based on treatment group and dose level, regardless of study phase, because the safety profile was expected to be generally uniform across tumor types.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 and Phase 2: INCB001158 50 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 mg BID starting on Day 1 of each 28-day cycle. In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and MSS-CRC (Phase 2) also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1 and Phase 2: INCB001158 75 mg + mFOLFOX6: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. In Phases 1 and 2, participants with advanced or solid metastatic tumors (Phase 1) and MSS-CRC (Phase 2) also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1 and Phase 2: INCB001158 100 mg + mFOLFOX6: In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and MSS-CRC (Phase 2) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous mFOLFOX6 (oxaliplatin 85 mg/m^2, leucovorin 400 mg/m^2, and 5-fluorouracil 400 mg/m^2 [bolus] and 2400 mg/m^2 [continuous infusion]) on Day 1 and Day 15 of each 28-day cycle after administration of INCB001158.
- Phase 1 and Phase 2: INCB001158 50 mg + Gemcitabine + Cisplatin: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle. In Phase 2, participants with BTC received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 25 mg/m^2 on Day 1 and 8 of each 28-day cycle, and participants with OC received intravenous gemcitabine 750 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and 8 of each 28-day cycle.
- Phase 1 and Phase 2: INCB001158 75 mg + Gemcitabine + Cisplatin: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. Participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle. In Phase 2, participants with BTC received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 25 mg/m^2 on Day 1 and 8 of each 28-day cycle, and participants with OC received intravenous gemcitabine 750 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and 8 of each 28-day cycle.
- Phase 1 and Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and with BTC or OC (Phase 2) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. In Phase 1, participants also received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and Day 8 of each 28-day cycle. In Phase 2, participants with BTC received intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 25 mg/m^2 on Day 1 and 8 of each 28-day cycle, and participants with OC received intravenous gemcitabine 750 mg/m^2 and intravenous cisplatin 30 mg/m^2 on Day 1 and 8 of each 28-day cycle.
- Phase 1 and Phase 2: INCB001158 50 mg + Paclitaxel: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50 mg BID starting on Day 1 of each 28-day cycle. In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and with GC, EC, or OC (Phase 2) received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 1 and Phase 2: INCB001158 75 mg + Paclitaxel: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 75 mg BID starting on Day 1 of each 28-day cycle. In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and with GC, EC, or OC (Phase 2) received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
- Phase 1 and Phase 2: INCB001158 100 mg + Paclitaxel: In Phases 1 and 2, participants with advanced or metastatic solid tumors (Phase 1) and GC, EC, or OC (Phase 2) received oral INCB001158 100 mg BID starting on Day 1 of each 28-day cycle. Participants with advanced or metastatic solid tumors (Phase 1) and with GC, EC, or OC (Phase 2) also received intravenous paclitaxel 80 mg/m^2 on Day 1, Day 8, and Day 15 of each 28-day cycle.
Arm/Group | Phase 1 and Phase 2: INCB001158 50 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 75 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 100 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 50 mg + Paclitaxel | Phase 1 and Phase 2: INCB001158 75 mg + Paclitaxel | Phase 1 and Phase 2: INCB001158 100 mg + Paclitaxel
Number analyzed (Participants) | 8 | 6 | 14 | 7 | 4 | 46 | 7 | 5 | 52
Participants | 8 | 6 | 13 | 7 | 4 | 46 | 7 | 5 | 51

2. Primary Outcome: Phase 1: Number of Participants With Any Dose-limiting Toxicity (DLT)
Description: A DLT was defined as the occurrence of any protocol-defined toxicity occurring up to and including Day 28, except those with a clear alternative explanation (e.g., disease progression) or transient (≤72 hours) abnormal laboratory values without associated clinically significant signs or symptoms based on investigator determination. All DLTs were assessed by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria.
Time Frame: up to Day 28
Population: Phase 1 DLT Evaluable Population: all participants enrolled in Phase 1 who had been treated with the assigned dose level of INCB001158 and who had received at least 32 of the 42 doses prescribed for a 21-day cycle regimen or at least 42 of the 56 doses prescribed for a 28-day cycle regimen (both representing ≥ 75% of the dose planned) or who had experienced a DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Recommended Phase 2 Dose (RP2D) of INCB001158 When Given in Combination With Each Chemotherapy Regimen
Description: The RP2D of the combination of INCB001158 and chemotherapy in 21-day (for gemcitabine/cisplatin) or 28-day (for mFOLFOX6 or paclitaxel) treatment cycles in participants with advanced or metastatic solid tumors was determined. After the dose escalation was completed, the INCB001158 dose level that was pharmacologically active and tolerable in combination with each chemotherapy regimen (i.e., maximum tolerated dose or lower) was determined to be the RP2D. The RP2D was then further assessed in tumor expansion cohorts in Phase 2.
Time Frame: up to Day 580
Population: DLT Evaluable Population
Measure: Number; unit: milligrams
Groups:
- All Phase 1 Participants: In Phase 1, participants with advanced or metastatic solid tumors received oral INCB001158 50, 75, or 100 mg BID plus intravenous modified FOLFOX6, intravenous gemcitabine 1000 mg/m^2 and intravenous cisplatin 30 mg/m^2, or intravenous paclitaxel 80 mg/m^2.
Arm/Group | All Phase 1 Participants
Number analyzed (Participants) | 54
milligrams | 100

4. Primary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), as determined by investigator assessment of radiographic disease as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Analysis was conducted by cohort (tumor type) in Phase 2 because different tumor types could have different response criteria or different background response rates.
Time Frame: up to 1385 days
Population: Phase 2 Response Evaluable Population: all participants who had received ≥1 dose of study treatment (INCB001158, mFOLFOX6, gemcitabine/cisplatin, or paclitaxel), completed a Baseline scan, and met ≥1 of the following criteria: (a) had ≥1 post-Baseline scan; (b) was in the study for a minimum of 63 days (8 weeks + 1 week window) of follow-up; (c) discontinued from study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 33 | 9 | 11 | 10 | 24
percentage of participants | 0.0 [0.0 to 36.9] | 24.2 [11.1 to 42.3] | 22.2 [2.8 to 60.0] | 9.1 [0.2 to 41.3] | 30.0 [6.7 to 65.2] | 16.7 [4.7 to 37.4]

5. Secondary Outcome: Phase 1: ORR
Description: ORR was defined as the percentage of participants with a confirmed best overall response of CR or PR, as determined by investigator assessment of radiographic disease as per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the Baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 580 days
Population: Phase 1 Response Evaluable Population: all participants who had received ≥1 dose of study treatment (INCB001158, mFOLFOX6, gemcitabine/cisplatin, or paclitaxel), completed a Baseline scan, and met ≥1 of the following criteria: (a) had ≥1 post-Baseline scan; (b) was in the study for a minimum of 63 days (8 weeks + 1 week window) of follow-up; (c) discontinued from study treatment. Analysis was conducted by dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7
percentage of participants | 12.5 [0.3 to 52.7] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 41.0] | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 60.2] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 52.2] | 28.6 [3.7 to 71.0]

6. Secondary Outcome: Phases 1 and 2: Duration of Response
Description: DOR was defined as the time from initial objective response (CR or PR) (as determined by investigator assessment of radiographic disease assessment per RECIST v1.1) until the earliest date of disease progression or death due to any cause, if it occurred sooner than disease progression. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 368 days
Population: Response Evaluable Population. Analysis was conducted based on study phase. Analysis was conducted by dose in Phase 1 and by cohort (tumor type) in Phase 2 because different tumor types could have different response criteria or different background response rates. Analysis was conducted in cohorts with >5 objective responders; the Kaplan Meier estimation method on a sample size of <5 responders is not valid. The confidence interval was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
months |  |  |  |  |  |  |  |  |  |  | 5.8 [4.1 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  |  |  |

7. Secondary Outcome: Phases 1 and 2: Disease Control Rate
Description: DCR was defined as the percentage of participants with an overall response of CR, PR, or stable disease (SD), as determined by investigator assessment of radiographic disease as per RECIST v1.1, for at least 8 weeks. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 1385 days
Population: Response Evaluable Population. Data analysis was conducted based on study phase. Additionally, analysis was conducted by dose in Phase 1 and by cohort (tumor type) in Phase 2 because different tumor types could have different response criteria or different background response rates.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7 | 8 | 33 | 9 | 11 | 10 | 24
percentage of participants | 62.5 [24.5 to 91.5] | 83.3 [35.9 to 99.6] | 16.7 [0.4 to 64.1] | 57.1 [18.4 to 90.1] | 75.0 [19.4 to 99.4] | 100.0 [39.8 to 100.0] | 42.9 [9.9 to 81.6] | 60.0 [14.7 to 94.7] | 85.7 [42.1 to 99.6] | 100.0 [63.1 to 100.0] | 66.7 [48.2 to 82.0] | 88.9 [51.8 to 99.7] | 54.5 [23.4 to 83.3] | 80.0 [44.4 to 97.5] | 66.7 [44.7 to 84.4]

8. Secondary Outcome: Phases 1 and 2: Progression-free Survival
Description: According to RECIST 1.1, PFS was defined as the length of time from the date of the first dose study of drug until the earliest date of disease progression, as determined by investigator assessment of radiographic disease per RECIST v1.1, or death due to any cause, if it occurred sooner than progression.
Time Frame: up to 1385 days
Population: FAS. Data analysis was conducted based on study phase. Additionally, analysis was conducted by dose in Phase 1 and by cohort (tumor type) in Phase 2 because different tumor types could have different response criteria or different background response rates. Median survival time was estimated using the Kaplan-Meier method. CI for median survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: INCB001158 50 mg + mFOLFOX6 | Phase 1: INCB001158 75 mg + mFOLFOX6 | Phase 1: INCB001158 100 mg + mFOLFOX6 | Phase 1: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1: INCB001158 50 mg + Paclitaxel | Phase 1: INCB001158 75 mg + Paclitaxel | Phase 1: INCB001158 100 mg + Paclitaxel | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 4 | 4 | 7 | 5 | 7 | 8 | 33 | 9 | 11 | 10 | 24
months | 3.7 [1.8 to 3.9] | 6.6 [1.7 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 1.7 [1.6 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 3.9 [0.6 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 5.3 [NA to NA] — The upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died. | 6.4 [3.7 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 3.9 [0.8 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 3.7 [1.5 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 11.8 [1.7 to 16.1] | 3.7 [2.8 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 8.5 [5.7 to 10.1] | 7.8 [2.2 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 3.5 [1.7 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 7.1 [3.5 to 11.1] | 3.7 [2.4 to 4.9]

9. Secondary Outcome: Cmin of INCB001158 in Participants Treated With INCB001158 in Combination With Chemotherapy on Cycle 2 Day 1 Following Repeated Dose Administration
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval. Extensive sample collection was used for the first 12 participants enrolled in each chemotherapy regimen. Sparse sample collection was used for the 13th participant enrolled and onward.
Time Frame: Day 1 of Cycle 2: predose; 0.5, 1, 2, 4, 6, and 8-10 hours post-dose for extensive sample collection. Day 1 of Cycle 2: predose; 1 and 4 hours post-dose for sparse sample collection
Population: Phase 2 Pharmacokinetic (PK) Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 7 | 17 | 8 | 8 | 5 | 13
nanograms per milliliter (ng/mL) | 747 (35.7) | 407 (407) | 268 (888) | 542 (102) | 1020 (27.2) | 633 (131)

10. Secondary Outcome: Cmax of INCB001158 in Participants Treated With INCB001158 in Combination With Chemotherapy Following the First Dose on Cycle 1 Day 1 and on Cycle 2 Day 1 Following Repeated Dose Administration
Description: Cmax was defined as the maximum observed plasma concentration over the dose interval. Extensive sample collection was used for the first 12 participants enrolled in each chemotherapy regimen. Sparse sample collection was used for the 13th participant enrolled and onward.
Time Frame: Day 1 of Cycles 1 and 2: predose; 0.5, 1, 2, 4, 6, and 8-10 hours post-dose for extensive sample collection. Day 1 of Cycles 1 and 2: predose; 1 and 4 hours post-dose for sparse sample collection
Population: Phase 2 PK Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 18 | 9 | 10 | 6 | 15
ng/mL
  Cycle 1 Day 1 | 1290 (16.4) | 1350 (35.2) | 2160 (22.3) | 1100 (68.0) | 1760 (17.2) | 1640 (23.2)
  Cycle 2 Day 1: number analyzed (Participants) | 7 | 17 | 8 | 8 | 5 | 13
  Cycle 2 Day 1 | 1960 (12.6) | 1860 (46.7) | 2250 (26.4) | 1600 (22.0) | 2390 (11.4) | 2100 (24.6)

11. Secondary Outcome: Tmax of INCB001158 in Participants Treated With INCB001158 in Combination With Chemotherapy Following the First Dose on Cycle 1 Day 1 and on Cycle 2 Day 1 Following Repeated Dose Administration
Description: tmax was defined as the time to the maximum concentration. Extensive sample collection was used for the first 12 participants enrolled in each chemotherapy regimen. Sparse sample collection was used for the 13th participant enrolled and onward.
Time Frame: as for outcome 10
Population: Phase 2 PK Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 18 | 9 | 10 | 6 | 15
hours
  Cycle 1 Day 1 | 4.13 [2.00 to 6.10] | 4.07 [1.97 to 7.53] | 4.08 [3.67 to 6.00] | 5.05 [2.25 to 7.50] | 4.09 [2.00 to 6.17] | 3.97 [1.78 to 6.08]
  Cycle 2 Day 1: number analyzed (Participants) | 7 | 17 | 8 | 8 | 5 | 13
  Cycle 2 Day 1 | 4.00 [1.80 to 7.50] | 4.00 [0.983 to 7.53] | 4.06 [2.03 to 6.02] | 4.13 [1.92 to 7.53] | 3.85 [3.77 to 3.92] | 3.95 [2.03 to 6.00]

12. Secondary Outcome: AUC0-t of INCB001158 in Participants Treated With INCB001158 in Combination With Chemotherapy Following the First Dose on Cycle 1 Day 1 and on Cycle 2 Day 1 Following Repeated Dose Administration
Description: AUC0-t was defined as the area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t. Extensive sample collection was used for the first 12 participants enrolled in each chemotherapy regimen. Sparse sample collection was used for the 13th participant enrolled and onward.
Time Frame: as for outcome 10
Population: Phase 2 PK Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x ng/mL
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 18 | 9 | 10 | 6 | 15
hours x ng/mL
  Cycle 1 Day 1 | 6910 (17.6) | 7240 (32.9) | 10600 (18.9) | 4680 (134) | 9290 (33.2) | 8840 (24.7)
  Cycle 2 Day 1: number analyzed (Participants) | 7 | 17 | 8 | 8 | 5 | 13
  Cycle 2 Day 1 | 11000 (21.1) | 10600 (55.3) | 12200 (34.4) | 10000 (18.4) | 14400 (13.7) | 12800 (30.3)

13. Secondary Outcome: Tlast of INCB001158 in Participants Treated With INCB001158 in Combination With Chemotherapy Following the First Dose on Cycle 1 Day 1 and on Cycle 2 Day 1 Following Repeated Dose Administration
Description: tlast was defined as the time of the last sample collected from which a concentration was measured. Extensive sample collection was used for the first 12 participants enrolled in each chemotherapy regimen. Sparse sample collection was used for the 13th participant enrolled and onward.
Time Frame: as for outcome 10
Population: Phase 2 PK Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: INCB001158 100 mg + mFOLFOX6: MSS-CRC (Cohort A1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: BTC (Cohort B1) | Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin: OC (Cohort B2) | Phase 2: INCB001158 100 mg + Paclitaxel: GC (Cohort C1) | Phase 2: INCB001158 100 mg + Paclitaxel: EC (Cohort C2) | Phase 2: INCB001158 100 mg + Paclitaxel: OC (Cohort C3)
Number analyzed (Participants) | 8 | 18 | 9 | 10 | 6 | 15
hours
  Cycle 1 Day 1 | 7.53 [7.47 to 8.00] | 7.73 [6.00 to 8.42] | 7.53 [7.50 to 8.05] | 7.50 [3.50 to 8.08] | 7.53 [7.50 to 7.67] | 7.65 [5.73 to 8.15]
  Cycle 2 Day 1: number analyzed (Participants) | 7 | 17 | 8 | 8 | 5 | 13
  Cycle 2 Day 1 | 7.50 [6.00 to 7.57] | 7.58 [7.50 to 8.38] | 7.60 [7.50 to 8.25] | 7.57 [7.50 to 8.00] | 7.55 [7.50 to 7.67] | 7.58 [7.48 to 8.25]

ADVERSE EVENTS:
Time Frame: up to 1385 days
Description: Treatment-emergent adverse events, defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug, have been reported. As pre-defined in the Statistical Analysis Plan, data analysis was conducted based on treatment group and dose level, regardless of study phase, because the safety profile was expected to be generally uniform across tumor types.
Groups:
- Total: Total
Arm/Group | Phase 1 and Phase 2: INCB001158 50 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 75 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 100 mg + mFOLFOX6 | Phase 1 and Phase 2: INCB001158 50 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 75 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin | Phase 1 and Phase 2: INCB001158 50 mg + Paclitaxel | Phase 1 and Phase 2: INCB001158 75 mg + Paclitaxel | Phase 1 and Phase 2: INCB001158 100 mg + Paclitaxel | Total
All-Cause Mortality (participants affected / at risk) | 4/8 | 2/6 | 11/14 | 4/7 | 3/4 | 30/46 | 5/7 | 4/5 | 36/52 | 99/149
Serious Adverse Events (participants affected / at risk) | 6/8 | 1/6 | 7/14 | 3/7 | 1/4 | 30/46 | 4/7 | 4/5 | 27/52 | 83/149
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 13/14 | 7/7 | 4/4 | 45/46 | 7/7 | 5/5 | 50/52 | 145/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 and Phase 2: INCB001158 50 mg + mFOLFOX6 (N=8) | Phase 1 and Phase 2: INCB001158 75 mg + mFOLFOX6 (N=6) | Phase 1 and Phase 2: INCB001158 100 mg + mFOLFOX6 (N=14) | Phase 1 and Phase 2: INCB001158 50 mg + Gemcitabine + Cisplatin (N=7) | Phase 1 and Phase 2: INCB001158 75 mg + Gemcitabine + Cisplatin (N=4) | Phase 1 and Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin (N=46) | Phase 1 and Phase 2: INCB001158 50 mg + Paclitaxel (N=7) | Phase 1 and Phase 2: INCB001158 75 mg + Paclitaxel (N=5) | Phase 1 and Phase 2: INCB001158 100 mg + Paclitaxel (N=52) | Total (N=149)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (2) | 9 (10)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (5) | 7 (10)
Assisted suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 6 (7)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 4 (6)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 7 (8)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 5 (6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 2 (3) | 9 (11)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 12 (12)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 and Phase 2: INCB001158 50 mg + mFOLFOX6 (N=8) | Phase 1 and Phase 2: INCB001158 75 mg + mFOLFOX6 (N=6) | Phase 1 and Phase 2: INCB001158 100 mg + mFOLFOX6 (N=14) | Phase 1 and Phase 2: INCB001158 50 mg + Gemcitabine + Cisplatin (N=7) | Phase 1 and Phase 2: INCB001158 75 mg + Gemcitabine + Cisplatin (N=4) | Phase 1 and Phase 2: INCB001158 100 mg + Gemcitabine + Cisplatin (N=46) | Phase 1 and Phase 2: INCB001158 50 mg + Paclitaxel (N=7) | Phase 1 and Phase 2: INCB001158 75 mg + Paclitaxel (N=5) | Phase 1 and Phase 2: INCB001158 100 mg + Paclitaxel (N=52) | Total (N=149)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 8 (11) | 14 (17)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (7) | 1 (1) | 1 (1) | 9 (18) | 1 (1) | 0 (0) | 15 (19) | 35 (50)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 5 (8) | 12 (15)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 4 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 9 (18) | 0 (0) | 0 (0) | 2 (2) | 14 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 18 (20) | 24 (26)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Amylase increased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (8) | 7 (13)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 25 (38) | 2 (3) | 1 (2) | 21 (30) | 64 (88)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 8 (10) | 0 (0) | 1 (1) | 11 (13) | 24 (28)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (5) | 1 (2) | 0 (0) | 4 (7) | 13 (18)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 9 (14) | 0 (0) | 0 (0) | 3 (4) | 16 (22)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 9 (14) | 1 (1) | 0 (0) | 9 (10) | 25 (33)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 6 (6) | 16 (17)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 13 (18) | 0 (0) | 0 (0) | 8 (9) | 26 (32)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 4 (8)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 3 (5) | 8 (11)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (3) | 2 (2) | 0 (0) | 2 (2) | 19 (29) | 1 (1) | 1 (1) | 13 (13) | 41 (53)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 2 (2) | 8 (10) | 27 (30)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 12 (14) | 2 (2) | 1 (1) | 10 (16) | 37 (45)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 9 (10) | 14 (18)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 3 (4) | 6 (7) | 2 (4) | 0 (0) | 11 (17) | 3 (3) | 1 (1) | 16 (25) | 45 (67)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 11 (13) | 2 (2) | 0 (0) | 10 (13) | 27 (33)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 6 (12) | 11 (17)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 9 (10)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 8 (9) | 4 (4) | 0 (0) | 7 (12) | 23 (29)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 5 (6)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 7 (10)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Fatigue (General disorders) | 3 (5) | 4 (4) | 4 (5) | 1 (1) | 1 (1) | 23 (33) | 2 (2) | 4 (5) | 29 (38) | 71 (94)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 9 (9)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 5 (6)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 10 (14) | 0 (0) | 0 (0) | 9 (9) | 22 (26)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (12) | 9 (13)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 5 (8) | 13 (23)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 4 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 9 (11)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 6 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 1 (1) | 1 (3) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 3 (3) | 14 (18)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 2 (3) | 0 (0) | 2 (2) | 13 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 8 (12) | 15 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 3 (3) | 11 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 5 (8) | 1 (2) | 0 (0) | 5 (9) | 16 (25)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 8 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 5 (5) | 15 (16)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (5)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (3) | 2 (2) | 3 (5) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 3 (6) | 12 (22)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 5 (6)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (5)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Mucosal ulceration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 1 (1) | 0 (0) | 5 (6) | 14 (17)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (6) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (9) | 12 (14)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 5 (6)
Nausea (Gastrointestinal disorders) | 5 (7) | 3 (6) | 5 (5) | 1 (1) | 1 (1) | 25 (44) | 3 (4) | 3 (3) | 21 (43) | 67 (114)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 6 (7) | 3 (3) | 0 (0) | 10 (12) | 22 (25)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 11 (25) | 0 (0) | 0 (0) | 7 (17) | 28 (52)
Neutrophil count decreased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 15 (31) | 0 (0) | 1 (1) | 9 (19) | 34 (62)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 9 (10) | 1 (1) | 1 (1) | 13 (20) | 29 (38)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 9 (10)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 10 (10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 9 (9)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (4) | 4 (4) | 0 (0) | 1 (1) | 6 (7) | 1 (1) | 2 (2) | 10 (11) | 27 (30)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 3 (4) | 2 (4) | 5 (9) | 0 (0) | 14 (29) | 0 (0) | 1 (1) | 3 (6) | 29 (54)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 6 (8) | 10 (14)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 9 (11) | 0 (0) | 2 (2) | 6 (8) | 23 (27)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 7 (7) | 14 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 6 (9) | 12 (16)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 10 (12) | 21 (23)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 6 (7)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 10 (16) | 0 (0) | 0 (0) | 1 (1) | 15 (22)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 10 (10)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 7 (9) | 17 (20)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 6 (15) | 13 (23)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 14 (26) | 1 (2) | 3 (6) | 18 (29) | 45 (72)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 12 (12)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
White blood cell count decreased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 8 (13) | 0 (0) | 0 (0) | 11 (28) | 28 (53)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03314935/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03314935/SAP_001.pdf